CLINICAL TRIAL: NCT02705378
Title: The Effect of Naloxegol on Refractory Constipation in the Intensive Care Unit
Acronym: NaRC-ICU
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI left institution. Protocol never submitted to the IRB, no contract executed only Confidentiality Agreement, and study not done.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NaRC-ICU_temp
Record Dates: First submitted 2016-02-05; First posted 2016-03-10 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Constipation; Critical Illness
Keywords: Intensive care unit; ICU; Critical Illness; Constipation
MeSH Terms: conditions — Constipation; Critical Illness | interventions — Polyethylene Glycols; polyethylene glycol 3350; naloxegol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Polyethylene glycol (Active Comparator): 17g power qday; reconstituted in water for naso/orogastric tube administration
  Interventions: Drug: Polyethylene glycol
- naloxegol (Experimental): 25mg qday; crushed pill reconstituted in water for naso/orogastric tube administration
  Interventions: Drug: naloxegol

INTERVENTIONS:
Drug: Polyethylene glycol — Intervention would be given by oro-gastric (OG) or naso-gastric (NG) tube
  Other Names: Polyethylene glycol (PEG); miralax; glycolax
  Arms: Polyethylene glycol
Drug: naloxegol — Intervention would be given by OG or NG tube
  Other Names: Movantik
  Arms: naloxegol

SUMMARY:
Naloxegol has recently been approved by the US Food and Drug Administration to treat opioid induced constipation in non-cancer chronic pain patients. Its effectiveness in acute care patients, however, is not known. Therefore, the researchers' goal is to investigate whether naloxegol is superior to osmotic laxatives for refractory constipation in ICU patients already receiving prophylactic stool softeners and simulant laxatives through a double-blind, randomized control trial.

DETAILED DESCRIPTION:
Constipation is often defined as the absence of a bowel movement for 3 consecutive days. The incidence of constipation in critically ill patients is estimated to be 50-80%. Constipation in the ICU is associated with various undesirable clinical outcomes, including: increased rate of infections, prolonged duration of mechanical ventilation, greater hospital length of stay, worsening of organ dysfunction, and even higher mortality.

Typical first-line agents for the management of ICU constipation include stool softeners (e.g. docusate) and bowel stimulants (e.g. senna glycol or bisacodyl), and these are often used prophylactically in critically ill patients. However, a significant proportion of patients require additional therapy to promote laxation , the most common being osmotic agents such as propylene glycol or lactulose. Often, multiple doses of osmotic agents over several days are required to achieve acceptable laxation rates during critical illness. As such, this has prompted the need for targeted therapy to improve constipation in the ICU.

Among major risk factors for constipation in the ICU are the lack of bowel stimulation via nutrition and exposure to high doses of continuous opioids . Indeed, clinical data suggests that early enteral nutrition promotes laxation in ICU patients. And recently, methylnaltrexone, a peripherally acting μ-opioid receptor antagonist, has shown promising results in its ability to reverse opioid-induced constipation. However, methylnaltrexone is delivered via subcutaneous injection and its absorption is likely to be variable in critically ill patients who often receive aggressive fluid resuscitation and have significant peripheral edema. The US Food and Drug Administration recently approved the use of naloxegol, a μ-opioid receptor antagonist available in tablet form, for the management of opioid-induced constipation in non-cancer chronic pain patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Admitted to an ICU at Massachusetts General Hospital (MGH)
3. Received ≥72 hours of continuous opioid infusion
4. Anticipated to require ≥48 hours of additional care in the ICU
5. Did not have a bowel movement in ≥72 hours
6. Allowed to receive (and tolerating) medications via nasogastric, orogastric, gastric, gastrojejunal, or oral route
7. Receiving at least trophic (10 mL/hr) of enteral nutrition

Exclusion Criteria:

1. Unable to provide informed consent or unavailable healthcare proxy
2. Not expected to survive >48 hours from time of enrollment
3. "Comfort measures only" status (i.e. palliative care)
4. Received medication other that docusate and senna glycoside for laxation
5. Had abdominal surgery that is expected to cause significant ileus
6. Mechanical bowel obstruction
7. Total bowel rest/exclusively receiving total parenteral nutrition
8. History of chronic constipation unrelated to opioid use
9. Compromised blood-brain-barrier
10. Current diagnosis of solid organ or hematologic cancer
11. On moderate/strong CYP3A4 inhibitors or strong CYP3A4 inducers
12. On other opioid antagonists
13. Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Laxation within 48 hours of starting second-line agent | From 72 hours after ICU admission until 120 hours after ICU admission
  Documented bowel movement (Yes/No) within 48 hours of randomization to receive second-line laxative agent

SECONDARY OUTCOMES:
Time to first bowel movement after starting second-line agent | From 72 hours after ICU admission until 120 hours after ICU admission
  Number of hours from initiation of a second-line laxative agent until first documented bowel movement
Doses of second-line laxative agent before bowel movement | From 72 hours after ICU admission until 120 hours after ICU admission
  Number of doses of second-line laxative agent until first documented bowel movement
Protein/caloric deficit | From admission to the ICU until the end of day 7 after ICU admission
  Cumulative calorie and protein deficits will be calculated in kcals and grams, respectively, utilizing standard clinical formulas from the day of ICU admission until day 7 of ICU admission
Feeding interruptions | From admission to the ICU until the end of day 7 after ICU admission
  Number of interruptions to enteral nutrition for high gastric residual volume during study period

CONTACTS AND LOCATIONS:
Overall Officials: Sadeq A. Quraishi, MD,MHA,MMSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patanwala AE, Abarca J, Huckleberry Y, Erstad BL. Pharmacologic management of constipation in the critically ill patient. Pharmacotherapy. 2006 Jul;26(7):896-902. doi: 10.1592/phco.26.7.896. PMID 16803421
- [Background] Mostafa SM, Bhandari S, Ritchie G, Gratton N, Wenstone R. Constipation and its implications in the critically ill patient. Br J Anaesth. 2003 Dec;91(6):815-9. doi: 10.1093/bja/aeg275. PMID 14633751
- [Background] van der Spoel JI, Oudemans-van Straaten HM, Kuiper MA, van Roon EN, Zandstra DF, van der Voort PH. Laxation of critically ill patients with lactulose or polyethylene glycol: a two-center randomized, double-blind, placebo-controlled trial. Crit Care Med. 2007 Dec;35(12):2726-31. doi: 10.1097/01.CCM.0000287526.08794.29. PMID 17893628
- [Background] Nassar AP Jr, da Silva FM, de Cleva R. Constipation in intensive care unit: incidence and risk factors. J Crit Care. 2009 Dec;24(4):630.e9-12. doi: 10.1016/j.jcrc.2009.03.007. Epub 2009 Jul 9. PMID 19592200
- [Background] Gacouin A, Camus C, Gros A, Isslame S, Marque S, Lavoue S, Chimot L, Donnio PY, Le Tulzo Y. Constipation in long-term ventilated patients: associated factors and impact on intensive care unit outcomes. Crit Care Med. 2010 Oct;38(10):1933-8. doi: 10.1097/CCM.0b013e3181eb9236. PMID 20639749
- [Background] van der Spoel JI, Schultz MJ, van der Voort PH, de Jonge E. Influence of severity of illness, medication and selective decontamination on defecation. Intensive Care Med. 2006 Jun;32(6):875-80. doi: 10.1007/s00134-006-0175-9. Epub 2006 Apr 28. PMID 16715327
- [Background] Reintam Blaser A, Poeze M, Malbrain ML, Bjorck M, Oudemans-van Straaten HM, Starkopf J; Gastro-Intestinal Failure Trial Group. Gastrointestinal symptoms during the first week of intensive care are associated with poor outcome: a prospective multicentre study. Intensive Care Med. 2013 May;39(5):899-909. doi: 10.1007/s00134-013-2831-1. Epub 2013 Jan 31. PMID 23370829
- [Background] Reintam A, Parm P, Kitus R, Starkopf J, Kern H. Gastrointestinal failure score in critically ill patients: a prospective observational study. Crit Care. 2008;12(4):R90. doi: 10.1186/cc6958. Epub 2008 Jul 14. PMID 18625051
- [Background] Herndon CM, Jackson KC 2nd, Hallin PA. Management of opioid-induced gastrointestinal effects in patients receiving palliative care. Pharmacotherapy. 2002 Feb;22(2):240-50. doi: 10.1592/phco.22.3.240.33552. PMID 11837561
- [Background] Masri Y, Abubaker J, Ahmed R. Prophylactic use of laxative for constipation in critically ill patients. Ann Thorac Med. 2010 Oct;5(4):228-31. doi: 10.4103/1817-1737.69113. PMID 20981183
- [Background] Azevedo RP, Freitas FG, Ferreira EM, Machado FR. Intestinal constipation in intensive care units. Rev Bras Ter Intensiva. 2009 Aug;21(3):324-31. English, Portuguese. PMID 25303556
- [Background] Sawh SB, Selvaraj IP, Danga A, Cotton AL, Moss J, Patel PB. Use of methylnaltrexone for the treatment of opioid-induced constipation in critical care patients. Mayo Clin Proc. 2012 Mar;87(3):255-9. doi: 10.1016/j.mayocp.2011.11.014. PMID 22386181
- [Background] Hewitt K, Lin H, Faraklas I, Morris S, Cochran A, Saffle J. Use of methylnaltrexone to induce laxation in acutely injured patients with burns and necrotizing soft-tissue infections. J Burn Care Res. 2014 Mar-Apr;35(2):e106-11. doi: 10.1097/BCR.0b013e31829b399d. PMID 23877147
- See also: Constipation in critically ill patients and its relationship to feeding and weaning from respiratory support — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3642590/